CLINICAL TRIAL: NCT05735743
Title: MoVE Trial: Motivational Strategies To Empower African Americans To Improve Dialysis Adherence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ebele Umeukeje, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 221538 - MoVE Trial; 1R01DK133530-01 (NIH)
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-04

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Dialysis treatment adherence; Hemodialysis; African Americans
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care
- Participants receiving intervention (Experimental): Motivational interviewing intervention
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — In this trial, motivational interviewing (MI) is the intervention. The MI sessions will embody the spirit of MI (PACE - Partnership, Acceptance, Compassion and Evocation) and the use of MI strategies (OARS - Open-ended questions, Affirmations, Reflections and Summaries) and MI communication processes (engagement, focusing, evoking and planning).
  Other Names: MI
  Arms: Participants receiving intervention

SUMMARY:
MoVE Trial is a randomized clinical trial designed to rigorously test the impact of a behavioral intervention (culturally tailored motivational interviewing - (MOVE)) delivered by trained health coaches, on hemodialysis treatment non-adherence. It is a a two-arm, parallel group randomized clinical trial with 24-week follow-up. It involves completion of surveys by patients enrolled in the study. It also involves participation in motivational interviewing sessions by patients who are randomized to the intervention (MI).

ELIGIBILITY:
Inclusion Criteria:

* African American
* Receiving hemodialysis treatments
* Been on hemodialysis for more than 30 days
* 18 years of age and older
* Within a 2-month look back at the time of screening, patients who have missed at least one dialysis session or shortened at least one dialysis session by 15 minutes.

Exclusion Criteria:

* Not self-identified as African American
* Impaired with mental status or severe illness
* Non-English speaking
* No documented evidence of dialysis treatment non-adherence
* Missed or shortened treatments due to hospitalizations or excused travel
* Terminal condition
* Living in a nursing home/rehab
* Planned transplant within the next 6 months
* Planned conversion to peritoneal dialysis within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Dialysis treatment adherence | Baseline to 24 weeks post-intervention
  Abstraction of dialysis treatment adherence data from the dialysis units' records which includes data on every treatment that occurred or should have occurred within the time frame. Records will reflect dialysis treatments which were completed, shortened, missed or did not occur due to hospitalizations, ER visits or travel.

SECONDARY OUTCOMES:
Change in Autonomous Regulation | Baseline, Week 8, Week 24
  Change in autonomous regulation will be measured by the 6-item Autonomous Regulation (AR) questionnaire. Questions range in score from 1 to 7, and overall score is a mean of all items (range 1 - 7). Lower scores reflect less autonomous regulation, and higher scores reflect greater autonomous regulation
Change in Autonomy Support | Baseline, Week 8, Week 24
  Change in autonomy support will be measured by the 6-item Health Care Climate (HCC) questionnaire. Questions range in score from 1 to 7, and overall score is a mean of all items (range 1 - 7). Lower scores reflect less autonomous support, and higher scores reflect greater autonomous support.
Change in Perceived competence | Baseline, Week 8, Week 24
  Change in perceived competence will be measured by the 8-item Perceived Kidney Disease Self-Management Scale (PKDSMS) questionnaire.Each question ranges in score from 1 to 5. Four of the items (#s 1, 2, 6, 7) are reversed-scored. The score is the sum of the 8 individual items. The total PKDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's (dialysis).
Change in Apathy | Baseline, Week 8, Week 24
  Change in apathy will be measured by the 7-item Apathy Evaluation Scale survey (AES-S) which measures three domains of apathy: deficits in goal-directed behavior; a decrement in goal-related thought content; and emotional indifference with flat affect. Each question ranges in score from 1 to 4. Item 3 is reverse-scored and then the sum of the 7 item scores is calculated. Range of scores is 7-28.
Change in Optimism | Baseline, Week 8, Week 24
  Change in optimism will be measured by the 10-item Life Orientation Test - Revised (LOT-R) questionnaire which assesses individual differences in generalized optimism versus pessimism. Only 6 of the 10 items on the revised LOT are used to derive an optimism score. Four of the items are filler items and are not used in scoring. Of the 6 survey questions utilized, each question ranges in score from 1 to 5. Thus, scores in principle can range from 6 to 30.

CONTACTS AND LOCATIONS:
Overall Officials: Ebele M Umeukeje, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (6):
- United States (6):
  - DaVita Philadelphia PMC Dialysis, Philadelphia, Pennsylvania
  - DaVita University City Dialysis, Philadelphia, Pennsylvania
  - Buttonwood DaVita Dialysis 449 N Broad St,, Philadelphia, PA 19123, Pennsylvania
  - Vanderbilt Dialysis Clinic, Nashville, Tennessee
  - Dialysis Clinic, Inc., Nashville, Tennessee
  - Vanderbilt Dialysis Clinic East, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No